CLINICAL TRIAL: NCT04564183
Title: Advancing Prevention of Pulmonary Fibrosis - A Cohort Study of Preclinical Pulmonary Fibrosis
Brief Title: Advancing Prevention of Pulmonary Fibrosis
Acronym: APPLe
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Mayo Clinic (Other); University of California, Los Angeles (Other); University of Texas (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1739
Record Dates: First submitted 2020-09-18; First posted 2020-09-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: IPF; Pulmonary Fibrosis; ILD
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Specimen Handling; Surveys and Questionnaires; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full Cohort: Entire study population
  Interventions: Other: Sample collection; Other: Questionnaires; Radiation: High resolution CT scan of the chest; Diagnostic Test: Pulmonary Function Test

INTERVENTIONS:
Other: Sample collection — Blood, Urine, Nail, Hair, Saliva, optional Stool
Other: Questionnaires — SF-36, Food Frequency, Pulmonary Fibrosis Study questionnaire, COVID questionnaire
Radiation: High resolution CT scan of the chest — Upon enrollment, all participants will undergo single prone volumetric thoracic chest CT scan. This will be performed at full inspiration using a 64-slice CT scanner.
Diagnostic Test: Pulmonary Function Test — All recruited participants will undergo a pre-bronchodilator spirometry test and a lung diffusion capacity test, both in accordance with ATS guidelines. Exercise capacity (maximum physical exertion) will be assessed by performing a 6-minute walk test, also according to ATS guidelines.

SUMMARY:
This study plans to learn more about pulmonary fibrosis and how it develops. We want to determine if the disease can be detected early, before the lung is permanently scarred.

This study will enroll participants who are not currently diagnosed with pulmonary fibrosis, but who have family members with pulmonary fibrosis. Because there is an increased risk within affected families, this cohort will allow us to learn how pulmonary fibrosis develops, and how the lungs change over time.

ELIGIBILITY:
Inclusion Criteria:

* Unaffected first degree relative from Familial Interstitial Pneumonia families (two or more family members with IIP)
* Age at least 40 years old and younger than 75 years old

Exclusion Criteria:

* Diagnosed with known (physician-diagnosed) pulmonary fibrosis prior to informed consent
* Other genetic diseases associated with interstitial lung disease
* Pregnant women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll up to 1,000 participants who are in families with two or more reported cases of pulmonary fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Screen all subjects for early Idiopathic Pulmonary Fibrosis (IPF) with High Resolution CT Scan of the Chest | Baseline
  All subjects will be screened with a high resolution CT scan to identify early signs of lung fibrosis. CT scans will be evaluated by study radiologists.

CONTACTS AND LOCATIONS:
Overall Officials: David Schwartz, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No